CLINICAL TRIAL: NCT04338035
Title: Fertility in Patients With Untreated Rectosigmoid Endometriosis
Brief Title: Fertility in Untreated Rectosigmoid Endometriosis
Status: Completed | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Principal Investigator, Fabio Barra, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: FERT-RECTOSIGM-ENDO
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Endometriosis; Bowel Endometriosis; Endometriosis, Rectum; Endometriosis Colon
MeSH Terms: conditions — Endometriosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rectosigmoid endometriosis
  Interventions: Behavioral: Expectant management

INTERVENTIONS:
Behavioral: Expectant management — Patients did not undergo surgical treatment for endometriosis and medical consultations were done every 6 months from the beginning of the attempts to conceive

SUMMARY:
Several studies investigated the reproductive outcomes after surgical treatment of colorectal endometriosis, mainly segmental colorectal resection. Little information is available on the spontaneous fertility of patients with bowel endometriosis. This study aims to evaluate the fertility of patients affected by rectosigmoid endometriosis who did not undergo previous surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Desire of conception
* Diagnosis of rectosigmoid endometriosis by transvaginal ultrasonography (TVS) and magnetic resonance imaging enema (MR-e)

Exclusion Criteria:

* Previous surgery for endometriosis
* Diagnosis of hydrosalpinx at imaging
* Previous conception
* Abnormal semen parameters of male partners

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with rectosigmoid endometriosis not undergoing surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 4-9 weeks after conception
  Ultrasonographic evidence of intrauterine gestational sac
Live birth rate | 22 weeks after conception
  Complete expulsion or extraction from a woman of a product of fertilization after 22 completed weeks of gestational age, which, after such separation, breathes or shows any other evidence of life

SECONDARY OUTCOMES:
Number (%) of patients conceiving spontaneously/by Assisted Reproductive Technology | Immediately after diagnosis of clinical pregnancy
  Modality of conception
Number (%) of patients undergoing vaginal delivery/delivering by cesarean section | 22-42 weeks after conception
  Modality of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Remorgida V, Ferrero S, Fulcheri E, Ragni N, Martin DC. Bowel endometriosis: presentation, diagnosis, and treatment. Obstet Gynecol Surv. 2007 Jul;62(7):461-70. doi: 10.1097/01.ogx.0000268688.55653.5c. PMID 17572918